CLINICAL TRIAL: NCT04459390
Title: Impact of Comorbidities on COVID19 Outcome
Brief Title: Association of Comorbidities With COVID19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebatallah Hassan, dr, Assiut University
Other Study IDs: COVID19
Record Dates: First submitted 2020-07-05; First posted 2020-07-07 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For initial diagnostic testing for SARS-CoV-2, CDC recommends collecting and testing an upper respiratory specimen. The following are acceptable specimens:
  * A nasopharyngeal (NP) specimen collected by a healthcare provider; or
  * An oropharyngeal (OP) specimen collected by a healthcare provider; or
  * Sputum specimen collected by a healthcare provider. Swab specimens should be collected using only swabs with a synthetic tip, and an aluminum or plastic shaft. Place swabs immediately into sterile tubes containing 2-3 mL of viral transport media. Store the samples at 2-8°C up to 72 hours. If a delay in shipping or extraction is expected, store samples at -70°C in accordance with CDC's protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19 with comorbidities: Patients with COVID19 with at least one of the following comorbidities:
  1. Hypertension
  2. Diabetes
  3. Cardiovascular disease
  4. Chronic pulmonary disease
  5. Obesity
  6. Chronic liver disease
  7. Chronic kidney disease
  8. Collagen vascular disease
  9. Autoimmune disease
  10. Malignancy
  Interventions: Diagnostic Test: realtime PCR
- COVID19 without comorbidities: Patients with COVID19 without any of the previously mentioned comorbidities
  Interventions: Diagnostic Test: realtime PCR

INTERVENTIONS:
Diagnostic Test: realtime PCR — Detection of SARS-CoV-2 genes by realtime PCR

SUMMARY:
Association of Comorbidities with unfavorable COVID19 outcomes as admission to intensive care, invasive ventilation or death.

DETAILED DESCRIPTION:
COVID19 is a new emerging, rapidly disseminating disease that consuming most of resources of efficient healthcare systems, and several hospitals, worldwide, are currently experiencing a shortage of ICU beds for critically ill patients with COVID-19 pneumonia.

A risk stratification based on clinical, radiological and laboratory parameters seems necessary in order to better identify those patients who may need hospital and/or ICU admission.

One of the most alarming clinical parameters in general is the presence comorbidities. The underlying diseases including hypertension, diabetes mellitus, respiratory system disease and cardiovascular disease, may be risk factors for severe COVID-19 patients with adverse outcomes compared with non-severe patients. Obesity is also a risk factor for COVID-19 severity with increased need to mechanical ventilation.

Chronic diseases share several features with infectious disorders, such as the proinflammatory state, and the attenuation of the innate immune response which may be linked etiologically to its pathogenesis.

Aim of the study:to assess the impact of comorbidities in patients with diagnosis of Covid-19 on outcome, in order to find the predictors of prolonged hospital stay, need for ICU admission or poor outcome

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Covid-19 test positive; hospitalized subjects; both sexes.

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population: Patients admitted to Assiut university Hospitals diagnosed as COVID19 positive patients by PCR. All patients will be subjected to full clinical assessment, some laboratory investigations which are potential marker of disease severity.
  Another studies include chest X ray and CT chest.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-10-20 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Rate of recovery/ ICU admission/ need for mechanical ventilation | Baseline
  The mean rate of recovery in patients with diagnosis of Covid19, who present with comorbidities at the time of hospital admission, with the mean recovery rate in patients without any of these comorbidities.
Time to improvement | Baseline
  Comparison of the survival curves (times to improvement) in the two groups (patients with and without comorbidities) and among patients presenting with different types of comorbidities.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang J, Zheng Y, Gou X, Pu K, Chen Z, Guo Q, Ji R, Wang H, Wang Y, Zhou Y. Prevalence of comorbidities and its effects in patients infected with SARS-CoV-2: a systematic review and meta-analysis. Int J Infect Dis. 2020 May;94:91-95. doi: 10.1016/j.ijid.2020.03.017. Epub 2020 Mar 12. PMID 32173574
- [Background] Simonnet A, Chetboun M, Poissy J, Raverdy V, Noulette J, Duhamel A, Labreuche J, Mathieu D, Pattou F, Jourdain M; LICORN and the Lille COVID-19 and Obesity study group. High Prevalence of Obesity in Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Requiring Invasive Mechanical Ventilation. Obesity (Silver Spring). 2020 Jul;28(7):1195-1199. doi: 10.1002/oby.22831. Epub 2020 Jun 10. PMID 32271993
- [Background] Badawi A, Ryoo SG. Prevalence of comorbidities in the Middle East respiratory syndrome coronavirus (MERS-CoV): a systematic review and meta-analysis. Int J Infect Dis. 2016 Aug;49:129-33. doi: 10.1016/j.ijid.2016.06.015. Epub 2016 Jun 21. PMID 27352628